CLINICAL TRIAL: NCT05117632
Title: An Open-label Study of ALTO-100 in Adults With Major Depressive Disorder and/or Post-traumatic Stress Disorder
Brief Title: ALTO-100 in MDD and/or PTSD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alto Neuroscience (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTO-100-001
Record Dates: First submitted 2021-11-02; First posted 2021-11-11 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Major Depressive Disorder; Post Traumatic Stress Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALTO-100 (Experimental): ALTO-100 PO tablet, daily dosing 8 weeks
  Interventions: Drug: ALTO-100 PO tablet

INTERVENTIONS:
Drug: ALTO-100 PO tablet — one tablet twice daily

SUMMARY:
The goal of this study is to collect biologically based data for defining predictors and correlates of the effects of ALTO-100.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of moderate to severe major depressive disorder (MDD) and/or post-traumatic stress disorder (PTSD)
* At baseline, either not taking an antidepressant medication, or currently taking a SSRI, SNRI, mirtazapine, or bupropion for at least 6 weeks with no dose modifications in the past 2 weeks
* Willing to comply with all study assessments and procedures
* Must not be pregnant or breastfeeding at time of enrollment or throughout study

Exclusion Criteria:

* Evidence of unstable cardiovascular, respiratory, liver, or renal impairment or disease
* Active suicidal ideation
* Diagnosed bipolar disorder, psychotic disorder, or dementia
* Current moderate or severe substance use disorder
* Has a history of hypersensitivity or allergic reaction to ALTO-100 or any of its components/excipients
* Concurrent or recent participation in another clinical trial for mental illness involving an investigational product or device

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
To understand the relationship between baseline biology and clinical outcome with ALTO-100 using the Montgomery-Åsberg Depression Rating Scale (MADRS) | Measured 5 times over 8 weeks
  The Montgomery-Åsberg Depression Rating Scale (MADRS) measures the severity of depression where smaller scores indicate less depression and higher scores suggest more severe depression. Possible scores for this 10 item version range from 0 to 60. The change from baseline to the end of the study is the primary outcome.
To understand the relationship between baseline biology and clinical outcome with ALTO-100 using the Clinical Global Impression scale - Severity (CGI-S) | Measured 5 times over 8 weeks
  The Clinical Global Impression scale - Severity (CGI-S) measures the severity of psychopathology in general where smaller scores indicate less illness and higher scores suggest more severe illness. Possible scores for this scale range from 1 to 7. The change from baseline to the end of the study is the primary outcome.
To understand the relationship between baseline biology and clinical outcome with ALTO-100 using the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | Measured 3 times over 8 weeks
  The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) measures the severity of PTSD where smaller scores indicate less severe PTSD and higher scores suggest more severe PTSD. Possible scores for this 30 item version range from 0 to 120. The change from baseline to the end of the study is the primary outcome.
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability of ALTO-100 | From the signing of the ICF until the follow-up visit (up to 12 weeks)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Number of Participants With Clinically Significant Vital Signs Abnormalities as a Measure of Safety and Tolerability of ALTO-100 | From the signing of the ICF until the end-of-treatment visit (up to 11 weeks)
  Vital signs measured include blood pressure, heart rate, respiratory rate, temperature, and weight.
Number of Participants With Clinically Significant Laboratory Abnormalities as a Measure of Safety and Tolerability of ALTO-100 | From the signing of the ICF until the end-of-treatment visit (up to 11 weeks)
  Blood samples for serum chemistry and hematology will be collected for clinical laboratory testing.

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Site 136, Tempe, Arizona
  - Site 139, Little Rock, Arkansas
  - Site 141, Costa Mesa, California
  - Site 118, Fresno, California
  - Site 116, Martinez, California
  - Site 116, Mather, California
  - Site 150, Boca Raton, Florida
  - Site 112, Doral, Florida
  - Site 155, Elgin, Illinois
  - Site 137, Noblesville, Indiana
  - Site 151, Baltimore, Maryland
  - Site 109, Belmont, Massachusetts
  - Site 108, Jackson, Mississippi
  - Site 142, Lincoln, Nebraska
  - Site 144, Las Vegas, Nevada
  - Site 146, Middleburg Heights, Ohio
  - Site 147, Fort Worth, Texas
  - Site 148, Fort Worth, Texas
  - Site 120, Houston, Texas
  - Site 113, Houston, Texas
  - Site 121, Draper, Utah
  - Site 105, Seattle, Washington
  - NTC Seattle (105a), Tacoma, Washington